CLINICAL TRIAL: NCT02849457
Title: Preventing Epilepsy Using Vigabatrin In Infants With Tuberous Sclerosis Complex (PREVeNT Trial) A Randomized, Double-blind, Placebo-controlled Seizure Prevention Clinical Trial for Infants With TSC
Brief Title: Preventing Epilepsy Using Vigabatrin In Infants With Tuberous Sclerosis Complex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Martina Bebin (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Martina Bebin, Professor of Neurology and Pediatrics, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PREVeNT; 1U01NS092595-01A1 (NIH)
Record Dates: First submitted 2016-07-13; First posted 2016-07-29 (Estimated); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-07

CONDITIONS: Tuberous Sclerosis Complex
MeSH Terms: conditions — Tuberous Sclerosis | interventions — Vigabatrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Delayed Vigabatrin (Placebo) (Placebo Comparator): Randomization will only occur after detection of epileptiform activity on EEG. Participants randomized to this arm will be treated with matching placebo until 24 months of age or until they show evidence of clinical seizures or electrographic seizures on video EEG. If electrographic or clinical seizures occur while on placebo, they will be eligible for Open label vigabatrin. Participants will be followed until 36 months of age.
  Interventions: Drug: Early Vigabatrin; Drug: Delayed Vigabatrin (Placebo)
- Early Vigabatrin (Experimental): Randomization will only occur after detection of epileptiform activity on EEG. Participants randomized to this arm will be treated with vigabatrin until 24 months of age or until they show evidence of clinical seizures or electrographic seizures on video EEG. If electrographic or clinical seizures occur while on vigabatrin, they will be eligible for Open label vigabatrin. Participants will be followed until 36 months of age.
  Interventions: Drug: Early Vigabatrin
- Watchful Waiting (Control Group) (No Intervention): Enrolled participants in this arm are those who never develop EEG abnormalities or clinical seizures during the length of the study. While all participants who enrolled in the study started in this group, participants were randomized upon development of EEG epileptiform activity. All participants who completed the study without developing EEG epileptiform activity or clinical seizures are reported in this group.

INTERVENTIONS:
Drug: Early Vigabatrin — Subjects randomized to vigabatrin will be treated with vigabatrin 100mg/kg/day until 24 months of age or until they show evidence of clinical seizures or electrographic seizures on video EEG. If electrographic or clinical seizures occur while on study drug, they will transition into the Open label phase of the study and continue to be followed until 36 months of age.
  Other Names: Sabril
  Arms: Delayed Vigabatrin (Placebo); Early Vigabatrin
Drug: Delayed Vigabatrin (Placebo) — Subjects randomized to placebo will be treated with matching placebo at 100mg/kg/day until 24 months of age or until they show evidence of clinical seizures or electrographic seizures on video EEG. If electrographic or clinical seizures occur while on study drug, they will transition into the Open label phase of the study and continue to be followed until 36 months of age.
  Arms: Delayed Vigabatrin (Placebo)

SUMMARY:
Study design is a Phase IIb prospective multi-center, randomized, placebo-controlled, double-blind clinical trial. The goal will be to enroll 80 infants with Tuberous Sclerosis Complex who are less than 6 months of age prior to the onset of their first seizure

DETAILED DESCRIPTION:
The central hypothesis of this Phase IIb trial is that early identification of electroencephalography (EEG) biomarkers and early treatment versus delayed treatment with vigabatrin in infants with tuberous sclerosis complex (TSC) will have a positive impact on developmental outcomes at 24 months of age. It would also prevent or lower the risk of developing infantile spasms and refractory seizures. This preventative approach would be expected to result in more favorable long-term cognitive, behavioral, developmental and psychiatric outcomes and significantly improve overall quality of life. It is a randomized, double-blind, placebo-controlled clinical trial design. Successful completion of this trial will also advance the field by demonstrating the value of systematic surveillance with EEG in asymptomatic infants with TSC.

ELIGIBILITY:
Inclusion Criteria:

1. less than or equal to 6 months of age
2. No history of seizures or infantile spasms, or evidence of subclinical electrographic seizures on a previous video EEG
3. Meet genetic or clinical diagnostic criteria for TSC, the latter based on current recommendations for diagnostic evaluation, such as physical exam, neuroimaging, echocardiogram

Exclusion Criteria:

1. Is greater than 6 months of age
2. Has not been diagnosed with TSC
3. History of seizures or infantile spasms, or evidence of subclinical electrographic seizures on a previous video EEG
4. Has received any anticonvulsant medication including vigabatrin, other anti-seizure therapeutic agent including cannabidiol
5. Has received an oral mTOR inhibitor such as everolimus or sirolimus
6. Has taken an investigational drug, including but not limited to cannabidiol, as part of a research study 30 days prior to enrollment, or plans on taking an investigational drug at any time during the duration of the study
7. Is currently enrolled, or plans on enrolling at any time during the duration of the study, in an experimental behavioral early intervention study
8. Has a history of being born prematurely (born less than <30 weeks gestation at the time of delivery)

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2016-12; Primary Completion 2023-04-26 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martina Bebin, MD, MPA, Principal Investigator — University of Alabama at Birmingham
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Boston Children's Hospital, Boston, Massachusetts
  - Beaumont Children's Hospital, Royal Oak, Michigan
  - Minnesota Epilepsy Group, PA, Saint Paul, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Cincinnati's Children Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with National Database for Autism Research (NDAR)

REFERENCES:
- [Result] Bebin EM, Peters JM, Porter BE, McPherson TO, O'Kelley S, Sahin M, Taub KS, Rajaraman R, Randle SC, McClintock WM, Koenig MK, Frost MD, Northrup HA, Werner K, Nolan DA, Wong M, Krefting JL, Biasini F, Peri K, Cutter G, Krueger DA; PREVeNT Study Group. Early Treatment with Vigabatrin Does Not Decrease Focal Seizures or Improve Cognition in Tuberous Sclerosis Complex: The PREVeNT Trial. Ann Neurol. 2023 Aug 28:10.1002/ana.26778. doi: 10.1002/ana.26778. Online ahead of print. PMID 37638552
- [Derived] van der Poest Clement E, Jansen FE, Braun KPJ, Peters JM. Update on Drug Management of Refractory Epilepsy in Tuberous Sclerosis Complex. Paediatr Drugs. 2020 Feb;22(1):73-84. doi: 10.1007/s40272-019-00376-0. PMID 31912454

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The PREVeNT clinical trial was conducted at 12 TSC Clinics in the U.S. with the first participant enrolled in December 2016 and last participant enrolled in March 2020. The study enrolled 84 TSC infants who were 6 months of age or younger and met the diagnostic criteria for TSC, with no history of seizures nor evidence of subclinical electrographic seizures on EEG. Participants were excluded if they were born prematurely, received any anti-seizure medication (ASM), or an mTOR inhibitor.
Groups:
- Delayed Vigabatrin (Placebo): Study drug (in this case, placebo) is given for administration, the entire content of one sachet (500 mg placebo) is dissolved in 10 ml water for oral administration that is dosed according to body weight 50-150 mg/kg/day divided BID. Dosing will follow established recommended guidelines (50 mg/kg/day and increased as needed by 50 mg/kg/day every 3 days up to a maximum dose of 150 mg/kg/day, divided BID).
  Participants randomized to this arm will be treated with matching placebo until 24 months of age or until they show evidence of clinical seizures or electrographic seizures on video EEG. If electrographic or clinical seizures occur while on placebo, they will be eligible for Open label vigabatrin. Participants will be followed until 36 months of age.
- Early Vigabatrin: Study drug (in this case, vigabatrin) is given for administration, the entire content of one sachet (500 mg vigabatrin) is dissolved in 10 ml water for oral administration that is dosed according to body weight 50-150 mg/kg/day divided BID. Dosing will follow established recommended guidelines (50 mg/kg/day and increased as needed by 50 mg/kg/day every 3 days up to a maximum dose of 150 mg/kg/day, divided BID).
  Participants randomized to this arm will be treated with vigabatrin until 24 months of age or until they show evidence of clinical seizures or electrographic seizures on video EEG. If electrographic or clinical seizures occur while on vigabatrin, they will be eligible for Open label vigabatrin. Participants will be followed until 36 months of age.
- Watchful Waiting (Open Label Vigabatrin): Participants in this group experienced seizures prior to detection of EEG epileptiform activity and where immediately placed on open label Vigabatrin.
Period: Enrolled, Pre-randomized Period
Arm/Group | Delayed Vigabatrin (Placebo) | Early Vigabatrin | Watchful Waiting (Control Group) | Watchful Waiting (Open Label Vigabatrin)
Started | 0 | 0 | 84 | 0
Completed | 0 | 0 | 72 | 0
Not Completed | 0 | 0 | 12 | 0
Not completed — Excluded prior to randomization due to discovery of exclusion criteria, e.g. prenatal mTOR inhibitor | 0 | 0 | 12 | 0
Period: Randomized Period
Arm/Group | Delayed Vigabatrin (Placebo) | Early Vigabatrin | Watchful Waiting (Control Group) | Watchful Waiting (Open Label Vigabatrin)
Started | 27 | 29 | 12 | 4
Completed | 22 | 29 | 11 | 4
Not Completed | 5 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Vigabatrin (Placebo) | Early Vigabatrin | Watchful Waiting (Control Group) | Total
Number analyzed (Participants) | 27 | 29 | 12 | 68
Age, Continuous [Mean (Standard Deviation); unit: Months] — Age at study enrollment
  Months | 1.9 (1.3) | 2.3 (1.4) | 4.4 (2.1) | 2.5 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 3 | 34
  Male | 12 | 13 | 9 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 5
  Not Hispanic or Latino | 23 | 28 | 10 | 61
  Unknown or Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Assessment Scores and Developmental Impact
Description: The primary outcome measure will be the standardized Cognitive scale scores on the Bayley Scales of Infant and Toddler Development- Third Edition at 24 months. The Cognitive scale Composite score is a standard score derived from the observed and elicited performance of the child on cognitive assessment tasks, with a mean of 100 and standard deviation of 10. The range for the Cognitive scale Composite score is 55 to 145. The score is calculated using standard procedures available in the manual for this measure. A higher score is considered better performance. The Bayley Scales of Infant and Toddler Development at 24 months will be used for the data analysis and to compare the developmental impact of early versus delayed treatment with vigabatrin.
Time Frame: 24 months
Population: The analysis population was the intent to treat population. Three participants withdrew prior to 24 months of age, and one participant did not complete the Bayley assessment at 24 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Vigabatrin (Placebo) | Early Vigabatrin | Watchful Waiting (Control Group) | Watchful Waiting (Open Label Vigabatrin)
Number analyzed (Participants) | 23 | 29 | 11 | 4
score on a scale | 83.9 (17.3) | 80.9 (15.6) | 97.3 (16.9) | 85.0 (21.6)
Statistical Analysis 1: Comparison: Delayed Vigabatrin (Placebo) vs Early Vigabatrin; Test type: Superiority; p = 0.8681, Mixed Models Analysis; Adjusted for age (<=7 vs >7 months) at randomization and sex. Unstructured covariance used among 12 and 24 month outcomes; Mean Difference (Final Values) = -0.6565, 95% CI 2-sided [-8.5567 to 7.2436], Standard Error of Mean 3.9332 — Parameter represents estimated amount difference in group means. Negative value represents higher mean in placebo group

2. Secondary Outcome: Number of Subjects That Develop Seizures When Treated With Study Drug During the Randomized Phase of the Study.
Description: Evaluate the number of subjects that develop seizures when treated with vigabatrin or placebo as a seizure prevention.
Time Frame: 24 months
Population: One participant in the Delayed Vigabatrin group withdrew prior to 24 months and prior to the development of any seizures. They were therefore excluded from count endpoints and from cognitive assessments at 24 months, although they were included in time to event analyses (censored at drop-out).
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Vigabatrin (Placebo) | Early Vigabatrin
Number analyzed (Participants) | 26 | 29
Participants | 19 | 20
Statistical Analysis 1: Comparison: Delayed Vigabatrin (Placebo) vs Early Vigabatrin; Test type: Superiority; p = 0.7375, Chi-squared

3. Secondary Outcome: Time to the Subject's First Clinical Seizure From Randomization
Description: Time to the subject's first clinical seizure will be measured for both subjects on placebo and vigabatrin.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: Months from randomization
Arm/Group | Delayed Vigabatrin (Placebo) | Early Vigabatrin
Number analyzed (Participants) | 27 | 29
Months from randomization | 2.77 [1.10 to 11.07] | 9.47 [4.80 to 22.27]
Statistical Analysis 1: Comparison: Delayed Vigabatrin (Placebo) vs Early Vigabatrin; Test type: Superiority; p = 0.1174, Regression, Cox; Adjusted for age (<=7 vs >7 months) at randomization and sex; Hazard Ratio (HR) = 0.593, 95% CI 2-sided [0.309 to 1.140]

4. Secondary Outcome: Count of Participants With Drug Resistant Epilepsy at 24 Months of Age.
Description: The count of participants with drug resistant epilepsy. Drug resistant epilepsy classified according to International League Against Epilepsy (ILAE) definition, specifically defined as any participant on 2 or more anti-seizure medications experiencing persistent seizures (seizures occurring within 3 months of the 24 month participant visit).
Time Frame: 24 months
Population: Three participants in the Delayed Vigabatrin group withdrew prior to age 24 months and could therefore not be classified as has having drug resistant epilepsy or not at age 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Vigabatrin (Placebo) | Early Vigabatrin
Number analyzed (Participants) | 24 | 29
Participants | 14 | 14
Statistical Analysis 1: Comparison: Delayed Vigabatrin (Placebo) vs Early Vigabatrin; Test type: Other — Two-sided test of non-equivalence; p = 0.4653, Chi-squared

5. Secondary Outcome: Evaluate Vineland II ABC Scores and Impact of Early Versus Late Treatment
Description: The range for the Vineland-II Adaptive Behavior Composite is 20 to 160
  The Vineland-II ABC standard score has a mean of 100 and standard deviation of 15, with higher scores indicating better overall adaptive functioning.
  The ABC standard score is a composite derived from obtained scores on the Communication, Daily Living Skills, Socialization, and Motor Skills domains on the Vineland-II and is calculated according to standardized procedures described in the Vineland-II manual.
Time Frame: 12 months, 24 months and 36 months
Population: The analysis population was the intent to treat population. Three participants withdrew prior to 24 months of age, and 2 withdrew prior to 12 months of age.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Vigabatrin (Placebo) | Early Vigabatrin | Watchful Waiting (Control Group) | Watchful Waiting (Open Label Vigabatrin)
Number analyzed (Participants) | 25 | 29 | 12 | 4
score on a scale
  12 months | 86.9 (13.1) | 86.0 (9.8) | 97.8 (14.2) | 86.3 (7.0)
  24 months: number analyzed (Participants) | 24 | 29 | 11 | 4
  24 months | 90.6 (14.3) | 84.9 (11.9) | 96.3 (5.8) | 85.3 (10.7)
  36 months: number analyzed (Participants) | 22 | 28 | 11 | 4
  36 months | 86.2 (17.5) | 78.6 (14.0) | 93.6 (8.8) | 76.8 (14.4)
Statistical Analysis 1: Comparison: Delayed Vigabatrin (Placebo) vs Early Vigabatrin; Test type: Superiority; p = 0.1697, Mixed Models Analysis; Adjusted for age at randomization (<=7 vs >7 months) and sex. Unstructured covariance used among 12, 24, and 36 month outcomes; Mean Difference (Final Values) = -4.4392, 95% CI 2-sided [-10.8346 to 1.9562], Standard Error of Mean 3.1889 — Pertains to the estimated difference in mean score between groups at study visit corresponding to 24 months of age

6. Secondary Outcome: Evaluate Autism Diagnostic Observation Schedule 2nd Edition (ADOS2) Scores and Impact of Early Versus Late Treatment
Description: Evaluate ADOS2 scores and the impact of early versus late treatment at 24 and 36 months.
Time Frame: 24 months and 36 months
Population: This outcome was not assessed because it required an in-person evaluation that could not be performed while wearing a face mask, which would have invalidated the assessment, and was thus eliminated as an outcome measure at the start of the COVID-19 pandemic.
Arm/Group | Delayed Vigabatrin (Placebo) | Early Vigabatrin | Watchful Waiting (Control Group) | Watchful Waiting (Open Label Vigabatrin)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects With Vigabatrin Related Adverse Events and Severe Adverse Events
Description: Number of subjects with vigabatrin related adverse events, severe adverse events as assessed by CTCAE v4.0 and risk evaluation and mitigation strategy (REMS) measures as required by the FDA.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Vigabatrin (Placebo) | Early Vigabatrin
Number analyzed (Participants) | 27 | 29
Participants | 6 | 2

8. Secondary Outcome: EEG Biomarker for Developing Epilepsy
Description: Feasibility of the routine 1 hour video EEG in determining the EEG biomarker for developing epilepsy. Outcome was determined as the number of participants developing seizures amongst those developing the biomarker (epileptiform activity).
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Vigabatrin (Placebo) | Early Vigabatrin | Watchful Waiting (Control Group) | Watchful Waiting (Open Label Vigabatrin)
Number analyzed (Participants) | 26 | 29 | 11 | 4
Participants | 19 | 20 | 0 | 4

ADVERSE EVENTS:
Time Frame: Adverse events occurring from enrollment through a patient's 36 month age visit (an average study duration of approximately 34 months). Note, patients could enroll at different ages, but had a common final study visit corresponding to age 36 months. Adverse events were assessed/collected at every study visit, and serious adverse events were collected in real time and reported to the medical safety monitor for the study.
Groups:
- Delayed Vigabatrin (Placebo), Pre-randomization: Patients who were eventually randomized to the Delayed Vigabatrin (Placebo) arm. The adverse events reflected in this arm occurred prior to randomization and initiation of study drug.
- Early Vigabatrin, Pre-randomization: Patients who were eventually randomized to the Early Vigabatrin arm. The adverse events reflected in this arm occurred prior to randomization and initiation of study drug.
- Delayed Vigabatrin (Placebo), Post-randomization: Study drug (in this case, placebo) is given for administration, the entire content of one sachet (500 mg placebo) is dissolved in 10 ml water for oral administration that is dosed according to body weight 50-150 mg/kg/day divided BID. Dosing will follow established recommended guidelines (50 mg/kg/day and increased as needed by 50 mg/kg/day every 3 days up to a maximum dose of 150 mg/kg/day, divided BID).
  Participants randomized to this arm will be treated with matching placebo until 24 months of age or until they show evidence of clinical seizures or electrographic seizures on video EEG. If electrographic or clinical seizures occur while on placebo, they will be eligible for Open label vigabatrin. Participants will be followed until 36 months of age.
- Early Post-randomization: Study drug (in this case, vigabatrin) is given for administration, the entire content of one sachet (500 mg vigabatrin) is dissolved in 10 ml water for oral administration that is dosed according to body weight 50-150 mg/kg/day divided BID. Dosing will follow established recommended guidelines (50 mg/kg/day and increased as needed by 50 mg/kg/day every 3 days up to a maximum dose of 150 mg/kg/day, divided BID).
  Participants randomized to this arm will be treated with vigabatrin until 24 months of age or until they show evidence of clinical seizures or electrographic seizures on video EEG. If electrographic or clinical seizures occur while on vigabatrin, they will be eligible for Open label vigabatrin. Participants will be followed until 36 months of age.
- Watchful Waiting (Open Label Vigabatrin), Before Use of Vigabatrin: Participants in this group eventually had a seizure and were placed on open label vigabatrin; however, the adverse events in this arm occurred prior to beginning open label vigabatrin.
- Watchful Waiting (Open Label Vigabatrin), After Starting Vigabatrin: Participants in this group experienced seizures prior to detection of EEG epileptiform activity and where immediately placed on open label Vigabatrin. The adverse events in this arm occurred after beginning open label vigabatrin.
Arm/Group | Delayed Vigabatrin (Placebo), Pre-randomization | Early Vigabatrin, Pre-randomization | Delayed Vigabatrin (Placebo), Post-randomization | Early Post-randomization | Watchful Waiting (Control Group) | Watchful Waiting (Open Label Vigabatrin), Before Use of Vigabatrin | Watchful Waiting (Open Label Vigabatrin), After Starting Vigabatrin
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29 | 0/27 | 0/29 | 0/12 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/27 | 2/29 | 14/27 | 15/29 | 1/12 | 2/4 | 2/4
Other Adverse Events (participants affected / at risk) | 4/27 | 4/29 | 15/27 | 17/29 | 7/12 | 3/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Vigabatrin (Placebo), Pre-randomization (N=27) | Early Vigabatrin, Pre-randomization (N=29) | Delayed Vigabatrin (Placebo), Post-randomization (N=27) | Early Post-randomization (N=29) | Watchful Waiting (Control Group) (N=12) | Watchful Waiting (Open Label Vigabatrin), Before Use of Vigabatrin (N=4) | Watchful Waiting (Open Label Vigabatrin), After Starting Vigabatrin (N=4)
Infections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders (Nervous system disorders) | 2 (2) | 0 (0) | 11 (30) | 10 (16) | 0 (0) | 2 (2) | 2 (2)
Cardiac disorders (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Vigabatrin (Placebo), Pre-randomization (N=27) | Early Vigabatrin, Pre-randomization (N=29) | Delayed Vigabatrin (Placebo), Post-randomization (N=27) | Early Post-randomization (N=29) | Watchful Waiting (Control Group) (N=12) | Watchful Waiting (Open Label Vigabatrin), Before Use of Vigabatrin (N=4) | Watchful Waiting (Open Label Vigabatrin), After Starting Vigabatrin (N=4)
Immune system disorders (Immune system disorders) | 1 (1) | 0 (0) | 3 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations (Infections and infestations) | 0 (0) | 2 (2) | 7 (30) | 8 (24) | 5 (9) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Investigations (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (5) | 7 (9) | 4 (7) | 1 (2) | 1 (2)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 4 (6) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 3 (4) | 3 (7) | 3 (3) | 0 (0) | 0 (0)
Eye disorders (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (5) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
General disorders (General disorders) | 2 (2) | 0 (0) | 3 (8) | 4 (11) | 0 (0) | 0 (0) | 1 (2)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
COVID-19 impacted one of the secondary endpoints (ADOS2) because of the requirement for facemasks during the assessment which would invalidate the ADOS2. Therefore this secondary outcome measure abandoned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT02849457/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT02849457/ICF_001.pdf